CLINICAL TRIAL: NCT04062448
Title: Phase 2 Study of Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib (PCI-32765) in Combination With Rituximab, in Japanese Patients With Waldenstrom's Macroglobulinemia (WM)
Brief Title: A Study of Ibrutinib in Combination With Rituximab, in Japanese Participants With Waldenstrom's Macroglobulinemia (WM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108666; 54179060WAL2002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib + Rituximab (Experimental): Participants will receive ibrutinib 420 milligram (mg) orally, once daily, from Day 1 of Week 1 until disease progression or unacceptable toxicity in combination with rituximab 375 milligram per square meter (mg/m^2) intravenously (IV) on Day 1 of Weeks 1 to 4 and Weeks 17 to 20.
  Interventions: Drug: Ibrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 420 mg will be administered orally.
  Other Names: PCI-32765
Drug: Rituximab — Rituximab 375 mg/m^2 will be administered intravenously.

SUMMARY:
The purpose of this study is to evaluate overall response rate (ORR) by Independent Review Committee (IRC) assessment, when combined with rituximab in Japanese participants with treatment naïve or relapsed/refractory Waldenstrom's Macroglobulinemia (WM).

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia (WM) in accordance with the consensus panel of the second International Workshop on Waldenstrom's Macroglobulinemia (IWWM)
* Japanese participants with treatment naïve or relapsed/refractory WM
* Measurable disease defined as serum monoclonal immunoglobulin M (IgM) greater than (>) 0.5 gram per deciliter (g/dL)
* Symptomatic disease, requiring treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (<=) 2
* Hematology and biochemical values within protocol-defined limits
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and agree to use highly effective methods of contraception while taking study drug. Women of childbearing potential must be practicing a highly effective, preferably user independent method of birth control during treatment with any drug in this study and for up to 12 months after the last dose of rituximab, 1 month after last dose of ibrutinib. Male participants must use an effective barrier method of contraception during the study and after receiving the last dose of ibrutinib, and for up to 12 months after last dose of rituximab if sexually active with a female of childbearing potential
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study. Participants must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Must be willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* Involvement of the central nervous system by WM
* Prior exposure to ibrutinib or other Bruton's Tyrosine Kinase (BTK) inhibitors
* Rituximab treatment within the last 12 months before the first dose of study intervention
* Received any WM-related therapy <=30 days prior to first administration of study treatment
* Plasmapheresis less than (<) 35 days prior to the initiation of study drug, except when at least one serum IgM central assessment was performed during the screening period and was >35 days from the most recent plasmapheresis procedure
* History of other malignancies
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Infection requiring systemic treatment that was completed <=14 days before the first dose of study drug
* Currently active, clinically significant Child-Pugh Class B or C hepatic impairment
* Inability or difficulty swallowing capsules, malabsorption syndrome, or any disease or medical condition significantly affecting gastrointestinal function
* Stroke or intracranial hemorrhage within 12 months prior to enrollment
* Currently active, clinically significant cardiovascular disease
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
* Infection with human immunodeficiency virus (HIV) or active infection with hepatitis B or hepatitis C virus
* Major surgery within 4 weeks of first dose of study drug
* Lactating or pregnant
* Male participants who plan to father a child while enrolled in this study or within 3 months after the last dose of ibrutinib, and within 12 months after last dose of rituximab
* Any contraindication to ibrutinib or rituximab including hypersensitivity to the active substance or to any of the excipients of ibrutinib or rituximab per local prescribing information
* Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before the planned first dose of study intervention or is currently enrolled in an investigational study
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg [for example], compromise the wellbeing) or that could prevent, limit, or confound the protocol-specified assessments
* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (9):
- Japan (9):
  - Kameda Medical Center, Chiba
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Nagoya City University Hospital, Nagoya
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka University Hospital, Suita
  - National Hospital Organization Disaster Medical Center, Tachikawa
  - University of Tsukuba Hospital, Tsukuba

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib + Rituximab: Treatment naive or relapsed/refractory Waldenstrom's Macroglobulinemia (WM) Japanese participants received ibrutinib 420 milligrams (mg) (3*140 mg capsules) orally, once daily, from Day 1 of Week 1 until disease progression or unacceptable toxicity along with rituximab 375 milligrams per square meter (mg/m^2) intravenously (IV) weekly for 4 consecutive weeks (Day 1 of Weeks 1 to 4), followed by a second course of once-weekly rituximab for 4 consecutive weeks (from Week 17 to 20) after a 12-week interval.
Period: Overall Study
Arm/Group | Ibrutinib + Rituximab
Started | 16
Completed | 13
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (11.21)
Age, Customized [Count of Participants; unit: Participants]
  Greater Than 65 | 11
  Less Than and Equal to (<=) 65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) According to the Modified Sixth International Workshop on Waldenstrom's Macroglobulinemia (IWWM) Criteria
Description: ORR is defined as the percentage of participants achieving a best overall response of confirmed complete response (CR), very good partial response (VGPR) or partial response (PR) according to the modified sixth IWWM criteria (National Comprehensive Cancer Network [NCCN] version 2, 2019), as assessed by the Independent Review Committee (IRC). CR: Immunoglobulin M (IgM) in normal range, disappearance of monoclonal protein by immunofixation, no histologic evidence of bone marrow involvement, resolution of any adenopathy/organomegaly (if present at baseline) along with no signs or symptoms attributable to Waldenstrom's Macroglobulinemia (WM); VGPR and PR: greater than or equal to (>=) 90 percent (%) (for VGPR) and >=50% (for PR) reduction of serum IgM, decrease in adenopathy/organomegaly (if present at baseline) on physical examination or computerized tomography (CT) scan, no new symptoms or signs of active disease.
Time Frame: Up to 1 year 11 months
Population: Response evaluable analysis set included all enrolled participants who had measurable disease at baseline, received at least 1 dose of ibrutinib and who had at least 1 adequate postbaseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 16
percentage of participants | 87.5

2. Secondary Outcome: Progression Free Survival (PFS) Assessed by Independent Review Committee
Description: PFS was defined as duration from the date of initial dose of ibrutinib to the date of first documented evidence of disease progression or death, whichever occurred first regardless of the use of subsequent antineoplastic therapy prior to documented disease progression or death. Kaplan-Meier method was used for the analysis.
Time Frame: From the date of initial dose up to 3 years and 5 months
Population: All treated analysis set included all enrolled participants who received at least 1 dose of ibrutinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 16
months | NA [NA to NA] — The median and 95% confidence interval were not estimable due to very less number of participants with events.

3. Secondary Outcome: Plasma Concentrations of Ibrutinib
Description: Plasma concentrations of ibrutinib were reported.
Time Frame: Day 1 of Week 4: Predose, 1 hour, 2 hours, 4 hours, and 6 hours postdose
Population: The Pharmacokinetic (PK) evaluable analysis set included all enrolled participants who had received at least 1 dose of ibrutinib and had at least 1 post-dose PK sample. Here, n (number analyzed) refers to number of participants evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 15
nanograms per milliliter (ng/mL)
  Week 4: Predose | 4.10 (6.15)
  Week 4: 1 hour postdose | 55.6 (74.6)
  Week 4: 2 hours postdose | 94.9 (147)
  Week 4: 4 hours postdose | 89.9 (115)
  Week 4: 6 hours postdose: number analyzed (Participants) | 14
  Week 4: 6 hours postdose | 50.5 (62.3)

4. Secondary Outcome: Plasma Concentrations of Metabolite PCI-45227
Description: Plasma concentrations of metabolite PCI-45227 were reported.
Time Frame: Day 1 of Week 4: Predose, 1 hour, 2 hours, 4 hours, and 6 hours postdose
Population: The PK evaluable analysis set included all enrolled participants who had received at least 1 dose of ibrutinib and had at least 1 post-dose PK sample. Here, n (number analyzed) refers to number of participants evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 15
ng/mL
  Week 4: Predose | 13.7 (14.8)
  Week 4: 1 hour postdose | 39.9 (42.3)
  Week 4: 2 hours postdose | 63.9 (62.3)
  Week 4: 4 hours postdose | 79.6 (51.5)
  Week 4: 6 hour postdose: number analyzed (Participants) | 14
  Week 4: 6 hour postdose | 65.6 (43.1)

5. Secondary Outcome: Number of Participants With Myeloid Differentiation Primary Response Gene 88 (MYD88) Biomarker Mutation
Description: Number of participants with MYD88 biomarker mutations were reported. MYD88 was assessed using next generation sequencing to detect the somatic mutations in the bone marrow aspiration samples collected during the study.
Time Frame: Day 1 of Week 1
Population: All treated analysis set included all enrolled participants who received at least 1 dose of ibrutinib. Here, 'N' (number of participants analyzed) refers to participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 7
Participants | 6

6. Secondary Outcome: Number of Participants With C-X-C Chemokine Receptor Type 4 (CXCR-4) Biomarker Mutations
Description: Number of participants with CXCR-4 biomarker mutations were reported. CXCR-4 was assessed using next generation sequencing to detect the somatic mutations in the bone marrow aspiration samples collected during the study.
Time Frame: Day 1 of Week 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 7
Participants | 2

7. Secondary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical event that occurred in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs were defined as any AE that occurred at or after the initial administration of study intervention through the day of last dose plus 30 days.
Time Frame: From first dose of study drug up to 30 days post last dose of study drug (that is, up to 40.6 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of ibrutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib + Rituximab
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: All-cause mortality: From Baseline (Day 1) up to 41 months; Serious and other events: From first dose of study drug up to 30 days after last dose of study treatment ((that is, up to 40.6 months)
Description: Safety analysis set included all enrolled participants who received at least 1 dose of ibrutinib. As ibrutinib and rituximab were administered as a combination treatment, adverse events analyses was not performed per the study intervention and thus combined data are presented.
Arm/Group | Ibrutinib + Rituximab
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 4/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib + Rituximab (N=16)
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Heat Illness (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthritis Bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 1
Escherichia Bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Heat Illness (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib + Rituximab (N=16)
Anaemia (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Supraventricular Extrasystoles (Cardiac disorders) | 1
Dry Eye (Eye disorders) | 2
Eyelid Oedema (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dental Caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1
Periodontal Disease (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Granuloma (General disorders) | 1
Malaise (General disorders) | 1
Oedema Peripheral (General disorders) | 2
Pyrexia (General disorders) | 4
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Acute Sinusitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Fungal Skin Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hepatitis B Reactivation (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Paronychia (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Pneumonia Fungal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 1
Blood Immunoglobulin A Decreased (Investigations) | 1
Blood Immunoglobulin G Decreased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 5
Platelet Count Decreased (Investigations) | 3
White Blood Cell Count Decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hypertonic Bladder (Renal and urinary disorders) | 1
Genital Rash (Reproductive system and breast disorders) | 1
Premenstrual Syndrome (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 2
Prostatomegaly (Reproductive system and breast disorders) | 1
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 2
Supraventricular Extrasystoles (Cardiac disorders) | 1
Dry Eye (Eye disorders) | 2
Eyelid Oedema (Eye disorders) | 1
Normal Tension Glaucoma (Eye disorders) | 1
Retinal Haemorrhage (Eye disorders) | 1
Abdominal Discomfort (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Anal Fissure (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dental Caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dry Mouth (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 2
Periodontal Disease (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Granuloma (General disorders) | 1
Malaise (General disorders) | 1
Oedema Peripheral (General disorders) | 2
Pyrexia (General disorders) | 5
Bile Duct Stone (Hepatobiliary disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Acute Sinusitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Fungal Skin Infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hepatitis B Reactivation (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Paronychia (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Pneumonia Fungal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 1
Blood Immunoglobulin A Decreased (Investigations) | 1
Blood Immunoglobulin G Decreased (Investigations) | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1
Liver Function Test Abnormal (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 5
Platelet Count Decreased (Investigations) | 3
White Blood Cell Count Decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Pancreatic Cystadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hypertonic Bladder (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Genital Rash (Reproductive system and breast disorders) | 1
Premenstrual Syndrome (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 2
Prostatomegaly (Reproductive system and breast disorders) | 1
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Umbilical Haemorrhage (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5
Internal Haemorrhage (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04062448/Prot_002.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT04062448/SAP_001.pdf